CLINICAL TRIAL: NCT00131287
Title: The Supplementary Effects of the Extract of Agaricus Blazei Murril on Type II Diabetes Mellitus (DM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ECbiotech Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH-EC-05-01
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Agaricus Blazei Murill; type II DM; insulin index
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Extract of Agaricus blazei Murill

SUMMARY:
The purpose of this study is to examine whether the extract of the Agaricus blazei Murill mushroom is effective in the supplementary treatment of type II DM patients.

DETAILED DESCRIPTION:
The researchers have the animal model that the extract of the Agaricus blazei Murill mushroom is effective in the treatment of type II DM mice conducted on 2002. The dose effects were also found. The researchers conducted the pilot study also showing the same effects in 2003. So the researchers designed this trial. The elixir of the Agaricus blazei Murill mushroom is popular in Taiwan for chronic diseases, such as type II DM.

ELIGIBILITY:
Inclusion Criteria:

* Type II DM
* Age 20-75 years old
* Treat with Gliclazide and Metformin
* Signed informed consent

Exclusion Criteria:

* GOT/GPT >80/80
* Creatinine > 2.0
* Lactating or pregnant women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108
Dates: Start 2005-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Percent reduction of glycated hemoglobin (HAb1C) and insulin resistance(HOMA-IR)

SECONDARY OUTCOMES:
Glucose, cholesterol, triglyceride, leptin, adiponectin comparisons

CONTACTS AND LOCATIONS:
Overall Officials: Hsu Chung-Hua, MD, Principal Investigator — Chinese Medicine Dep, Taipei Hospital
Locations (1):
- Chung-Hua Hsu, Taipei, Taiwan